CLINICAL TRIAL: NCT02686320
Title: Prospective Study of Evolution of Rheumatoid Arthritis After 65 Years Old
Brief Title: Prospective Study of Patients With Rheumatoid Arthritis After the Age of 65
Acronym: PRESAGE
Status: Terminated | Type: Observational
Why Stopped: Study suspended due to lack of PI to handle it
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Other Study IDs: NI-2015
Record Dates: First submitted 2016-02-05; First posted 2016-02-19 (Estimated); Last update posted 2025-11-20 (Actual); Status verified 2025-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Rheumatoid arthritis; Elderly; infections; cardio-vascular disease; osteoporosis; cancer
MeSH Terms: conditions — Arthritis, Rheumatoid; Infections; Osteoporosis; Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Rheumatoid arthritis >65 years old
- Rheumatoid arthritis <50 years old

SUMMARY:
Rheumatoid arthritis (RA) is associated with a higher prevalence of infections, malignancies, osteoporotic fractures and cardiovascular diseases. Few data are available regarding the prevalence and severity of these comorbidities in elderly RA patients. The purpose of this study is to determine the effect of age on prevalence and severity of comorbidities in RA.

DETAILED DESCRIPTION:
Prevalence of rheumatoid arthritis (RA) in elderly is increasing because of the increasing life expectancy. RA is associated with a higher prevalence of infections, malignancies, osteoporotic fractures and cardiovascular diseases. The purpose of this study is to determine the effect of age on prevalence and severity of comorbidities in RA. This study also aims to determine whether age influences disease progression and efficacy and tolerance of treatments.

This study will compare two groups of patients : patients older than 65 years old and patients younger than 50 years old, matched for gender and disease duration.

The first part of the study will be cross-sectional and will aim to compare characteristics regarding RA manifestations and comorbidities of the two groups at inclusion.

Whereas the second part will be prospective to assess the occurrence of comorbidities and the efficacy and safety of treatments in these two groups. Patients will be assessed every year during 5 years in accordance with usual follow-up of the patients.

This study could help to better manage elderly RA patients and to modify clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Rheumatoid arthritis according to American College of Rheumatology (ACR) /Eular 2010 criteria or American College of Rheumatalogy 1987 criteria
* Age >65 years or patients between 18 and 50 years matched for sex and disease duration with the group of elderly patients (control group)

Exclusion Criteria:

* Patients who do not understand rules and implications of the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Rheumatoid arthritis patients from department A and B of rheumatology in Cochin hospital
Sampling Method: Non-Probability Sample
Enrollment: 176 (Actual)
Dates: Start 2016-03-29 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-05-30 (Actual)

PRIMARY OUTCOMES:
Number of severe infections | 5 years
  Occurrence of severe infection requiring hospitalization or varicella-zoster virus
Number of cancers | 5 years
  Occurrence of solid cancer or hemopathy
Number of cardiovascular diseases | 5 years
  Occurrence of myocardial infarction or stroke
Number of osteoporotic fractures | 5 years

SECONDARY OUTCOMES:
Disease Activity Score (DAS 28) | 5 years
  to evaluate articular activity
Simple Disease Activity Index (SDAI) | 5 years
  to evaluate clinical articular activity of rheumatoid arthritis
Erythrocyte sedimentation rate | 5 years
  to evaluate biological articular activity of rheumatoid arthritis
Measure of C-reactive protein (CRP) | 5 years
  to evaluate biological articular activity of rheumatoid arthritis
Number of synovitis and/or tenosynovitis at ultrasound of hands | 5 years
  to evaluate articular activity of rheumatoid arthritis at ultrasound
Health assessment questionnaire (HAQ) score | 5 years
Need of orthopaedic surgery | 5 years
  to evaluate severity of rheumatoid arthritis
Number of erosions at X-rays (hands and feet) | 5 years
  to evaluate severity of rheumatoid arthritis
Number of diabetes, arterial hypertension and dyslipidaemia | 5 years
  to evaluate risks factor of cardiovascular disease
Number of cataracts | 5 years
Number of vaccinations | 5 years
  Previous influenza vaccination within the previous year and pneumococcal vaccination within the previous 5 years will be searched during medical interview.

CONTACTS AND LOCATIONS:
Overall Officials: Yannick ALLANORE, MD, PhD, Principal Investigator — Assistance Publique- Hôpitaux de Paris, Cochin Hospital
Locations (1):
- Cochin hospital, Paris, Paris, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Soubrier M, Tatar Z, Couderc M, Mathieu S, Dubost JJ. Rheumatoid arthritis in the elderly in the era of tight control. Drugs Aging. 2013 Nov;30(11):863-9. doi: 10.1007/s40266-013-0122-8. PMID 24105334
- [Background] Widdifield J, Bernatsky S, Paterson JM, Gunraj N, Thorne JC, Pope J, Cividino A, Bombardier C. Serious infections in a population-based cohort of 86,039 seniors with rheumatoid arthritis. Arthritis Care Res (Hoboken). 2013 Mar;65(3):353-61. doi: 10.1002/acr.21812. PMID 22833532